CLINICAL TRIAL: NCT05377099
Title: Evaluation of the Change in the Deformation Amplitude Ratio, Integrated Radius and Stress Strain Index as Parameters of Corneal Biomechanics Post Different Laser Vision Correction Procedures
Brief Title: Evaluation of the Change in the DA Ratio, IR and SSI as Parameters of Corneal Biomechanics Post Different LVC Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wessam Salem, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD 187-2020
Record Dates: First submitted 2022-05-01; First posted 2022-05-17 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Corneal Biomechanics
Keywords: CORVIS - Corneal Biomechanics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser In situ Keratomileusis (LASIK) (Active Comparator): Measurement of the deformation amplitude ratio, integrated radius and stress strain index as corneal biomechanical indices in refractive patients before and after LASIK
  Interventions: Diagnostic Test: CORVIS
- Femto-second assisted LASIK (FS-LASIK) (Active Comparator): Measurement of the deformation amplitude ratio, integrated radius and stress strain index as corneal biomechanical indices in refractive patients before and after Femto LASIK
  Interventions: Diagnostic Test: CORVIS
- Photorefractive Keratectomy (PRK) (Active Comparator): Measurement of the deformation amplitude ratio, integrated radius and stress strain index as corneal biomechanical indices in refractive patients before and after PRK
  Interventions: Diagnostic Test: CORVIS

INTERVENTIONS:
Diagnostic Test: CORVIS — Measurement of the DA ratio, IR and SSI before and after for patients under gone LASIK, femto LASIK and PRK using the CORVIS device.

SUMMARY:
In the study, The Investigators will compare the participates' corneal biomechanical properties including:

Deformation Amplitude ratio (Da Ratio) Integrated Radius (IR) Stress strain index (SSI)

All measurements will be taken before and after 3 months of LVC.

DETAILED DESCRIPTION:
Each Participant will undergo preoperative pentacam and corvis scan for his eyes and the 3 months post operative.

The participants are divided into 3 groups, one who underwent LASIK, one PRK and one Femto LASIK.

Collected data will before and after surgery will be compared in each arm and then the 3 arms will be compared together.

ELIGIBILITY:
Inclusion Criteria:

* • Age range 18 - 40 years.

  * Normal eyes with normal tomographic indices.
  * Patients with maximum mean refractive spherical equivalent (MRSE) of -7.00 diopters and with maximum astigmatism of -3.00 diopters.

Exclusion Criteria:

* • Patients with any other coexisting corneal diseases.

  * Keratoconus eyes.
  * Eyes with previous refractive corneal surgery.
  * Patients with increased intraocular pressure.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the changes in DA ratio, integrated radius and SSI before and after LVC | 3-6 months post operative
  Comparison between in DA ratio (DA ratio) in patients undergoing LASIK, Femto LASIK and PRK.
  Comparison between changes in integrated Radius (IR) in patients undergoing LASIK, Femto LASIK and PRK.
  Comparison between changes in Stress strain index (SSI) in patients undergoing LASIK, Femto LASIK and PRK.
  Each indices will be compared before and after the Laser vision correction (LVC) procedure and the indices are not to be compared to each other to have have a fixed unit measure.
  I reviewed your comment and I dont see any conflicts, to clarify how multiple measurements will be aggregated to arrive at one reported value again I am going to measure each index and compare it with "itself' before and after 3 different LVC.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hosny, Principal Investigator — Cairo University; Mohamed Anis, Study Director — Cairo University; Wessam Salem, Study Chair — Cairo University; Mohamed ELnaggar, Study Director — Research institute of Ophthalmology
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No